CLINICAL TRIAL: NCT01796639
Title: Retrospective Study of Long-term Survival and Related Factors Among Kidney Transplant Recipients in China
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: COLO400ACN02
Record Dates: First submitted 2013-02-16; First posted 2013-02-22 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- kidney transplantation patients with living-donor grafts

SUMMARY:
The primary objective of this study is to evaluate graft survival and recipient survival among kidney transplant recipients in China, and also to analyze possible factors related to patient and graft survival.

The secondary objective is to evaluate several secondary outcomes among kidney transplant recipients, such as average creatinine value, acute rejection episodes, NODM, incidence of BKV infection etc. At the same time analyze possible impact factors related to these secondary outcomes.

DETAILED DESCRIPTION:
Renal transplantation is the choice for patients with end-stage renal disease. In the past two decades, progress in surgical procedure, medical care, and immunosuppression have significantly improved the short-term results of organ transplantation. Nevertheless, grafts continue to fail over time, these improvements in immunosuppression and reduced incidence of acute rejection episodes have had only minimal effects on chronic allograft dysfunction and late graft loss. Long-term patient's death and graft failure are the main limitations for a better performance of renal transplant programs.

Multiple factors have been shown to affect the outcome of renal transplantation. These include demographic characteristics such as race and ethnicity, pretransplantation dialysis course, the timing of the transplantation，and the patients' co morbidities. Patient response to the transplantation procedure (e.g., delayed graft function, acute rejection, and acute tubular necrosis) is strongly associated with the long-term prognosis. In the last decade, with the increase of immunosuppressive agents in our therapeutic arsenal, several attempts have been made to improve graft performance. However, the majority of trials aiming to avoid calcineurin inhibitor (CNI)-related nephrotoxicity only reported short-term data. Also, and because of the lack of assessment of the role of the different ethiopathogenic factors that lead to graft damage, just avoiding CNI-related nephrotoxicity may be an oversimplification of the problem in the prevention of graft attrition.

There are many studies which have evaluated the long-term outcomes of graft and patient survival and have analyzed multiple relative factors. Unfortunately, such data in Chinese population are lacking. Meanwhile, the situation in China is somewhat different with others, such as race, the dosage of immunosuppressant and so on. A better characterization of the weight of immune and non-immune factors responsible for graft damage may help us to improve the outcomes in transplant recipients. Studies derived from well-designed and well-performed patient registries can provide a real world view of clinical practice, patient outcomes, safety, and comparative effectiveness and cost effectiveness. The goal of this project is to analyze retrospective data collected by disease registry, then to evaluate the graft and recipient outcomes of kidney transplants and relative impact factors.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* Received a transplant from Jan 1,1995 to Dec 31, 2007, only including those with living donor grafts
* Age: 18-75 years

Exclusion Criteria:

* Multiple-organ transplant recipients
* Patients records with missing information in 12 months post-transplantation
* Patients who did not have the information regarding their maintenance immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female kidney transplantation patients with living-donor grafts, > 18 years of age
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Graft survival | 5-year
  Graft survival, measured as the time between kidney transplant and the failure of the graft.
Recipient survival | 5-year
  measured as the time between the most recent kidney transplant and the patient's death. Graft outcome was censored at the earliest of the following events and was analyzed as days to graft failure or censor: loss to follow-up, patient death.

SECONDARY OUTCOMES:
Average creatinine value | 5 years
The rate of acute rejection episodes | 5 years
The incidence of BPAR and its severity | 5 years
The incidence of NODM | 5 years
The incidence of infection | 5 years
The incidence of biopsy proven CNIs nephrotoxicity | 5 years
The rate of posttransplantation malignancies | 5 years

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - The 309th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - The First affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shenyang Military General Hospital, Shenyang, Liaoning
  - Jinan Military General Hospital, Jinan, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Medical College of Xian Jiaotong University, Xian, Shanxi
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang